CLINICAL TRIAL: NCT00172120
Title: An 18-month, Open-label Extension Study of Once-daily ALX1-11 for the Treatment of Postmenopausal Women With Osteoporosis (TRES)
Brief Title: Open Label Extension
Acronym: TRES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-11-016
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Post-menopausal; Osteoporosis; Parathyroid Hormone; PTH; ALX1-11
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALX1-11

SUMMARY:
TRES will evaluate the effects of continued ALX1-11 treatment on the safety and efficacy variables assessed in the OLE study for a maximum treatment duration of 36 months in OLES and TRES combined.

DETAILED DESCRIPTION:
The primary goal of osteoporosis therapy is to prevent fracture, and anabolic agents can accomplish this by strengthening bone structure, which is accompanied by changes in BMD. Effects of ALX1-11 on BMD have been previously documented in a dose-finding Phase II clinical trial in osteoporotic postmenopausal women taking calcium and vitamin D supplements, who were otherwise naive to osteoporosis therapies. The anabolic effects of ALX1-11 on lumbar vertebrae were statistically significant compared to placebo after 12 months of treatment. In addition, animal studies showed that the new bone formed by treatment with ALX1 11 is of good quality both histologically and biomechanically (Mosekilde et al., 1991; Kimmel et al., 1993).

Protocol ALX1-11-93001 (TOP) assessed the effect of 18 months of ALX1-11 treatment on fracture incidence as a primary efficacy variable, and Protocol CL1-11-002 (OLES) assessed the effect on BMD for up to 24 months of treatment. Subjects who will be enrolled in the current study (TRES) will be those who received placebo in TOP and ALX1-11 in OLES. TRES will evaluate the effects of continued ALX1-11 treatment on the safety and efficacy variables assessed in the OLE study for a maximum treatment duration of 36 months in the OLES and TRES combined.

ELIGIBILITY:
Inclusion Criteria:

* Received placebo in TOP
* Completed 18 months of daily treatment with ALX1-11 in OLES
* Received their last dose of ALX1-11 in OLES within 3 months (90 days) of dosing in this study
* Have the ability to continue to self-administer, or have a designee administer, a daily injection
* Have the ability to understand, and willingness to sign, an informed consent form (ICF)

Exclusion Criteria:

Subjects are excluded who have developed any of the exclusion criteria for OLES, or modifications as listed below.

Concurrent Diseases Subjects are excluded if they have developed any of the diseases or illnesses listed since enrollment in OLES.

* Immune.Significant* immunological disorders; including AIDSAllergies to ALX1-11 or its constituents
* Endocrine.Significant* endocrine disorders, including hyper or hypoparathyroidism, Cushing's disease, hyperthyroidism
* Gastrointestinal (GI).Significant* GI disorders
* Kidney and Collecting.Significant* renal disorders or impaired renal function, nephrolithiasis or urolithiasis, verified kidney calcification, etc.
* Liver, biliary tract, pancreatic.Significant* hepatic or pancreatic disorders, active hepatitis, or pancreatitis
* Musculoskeletal.Metabolic bone disease, eg., Paget's disease, osteogenesis imperfecta, or osteomalacia -Chronic, active joint disease and/or joint infection
* Neoplasia.Cancer, with the exception of squamous or basal cell carcinoma**
* Nervous.Significant* neurological or psychiatric disease
* Vascular, respiratory, and cardiac.Significant* unstable cardiac or pulmonary disease

(*)Significance will be determined by the investigator on the basis of history, physical exam, and/or laboratory screens. Significant disorders necessitate ongoing changes in therapeutic medication or frequent monitoring.

(**)Subjects who have had either squamous or basal cell carcinoma of the skin can enroll if: 1. The lesion(s) was fully resected with clear margins described in a written report by a pathologist, AND 2. The subject has had no recurrence of lesions for at least 1 year from the time of the original resection

Prohibited Concomitant Medications

* PTH analogs*
* Fluoride
* Strontium
* Calcitonin
* Vitamin D metabolites or analogs(eg., calcitriol)
* Immunomodulatory agents with antiproliferative activity
* Cytostatics**
* Thyroxine. Prohibited if dose > 0.2 mg/day (see Table 4-4 for allowed conditions)
* Bisphosphonate
* Anabolic steroids or androgens

(*)PTH (parathyroid hormone) analogs include PTH(1-34), PTHrP, and other analogs

(**)eg, azathioprine, recombinant human tumor necrosis fusion (Fc) protein, monoclonal antibody against tumor necrosis factor (e.g., infliximab [Remicade™])

Medications Requiring a Washout Period - Subjects who completed OLES and then began taking medications listed in the following table may enroll in this study after a washout period of 30 days.

* Hormone-replacement therapy*
* Methotrexate
* SERMs**
* Any investigational drug
* Other medications known to affect the metabolism of bone
* 30 days with PMO approval

(*)Includes estrogen- and estrogen/progesterone-replacement therapy given by oral, transdermal, or intramuscular administration b SERMs (selective estrogen receptor modulator) include tamoxifen and raloxifene (Evista®) PMO = project medical officer

(**)SERMs (selective estrogen receptor modulator) include tamoxifen and raloxifene (Evista®) PMO = project medical officer

Medications Allowed if Specific Conditions Are Met-Medications that are allowed under specific conditions are listed:

* Thyroid hormone. At a stable dose <= 0.2 mg/day
* Thiazide. At a stable dose
* Vaginal application of estrogen-containing creams. Conjugated estrogen or estradiol at a dose of <=0.5 g administered twice each week (total of 1.0 g weekly). Estrace® (Ogen)at a dose <=1.0 g twice each week (total of 2.0 g weekly)
* Systemic corticosteroids. Acute bolus of steroids (oral or injectable) for a self-limited illness allowed under the following conditions: 1. Exposure to steroids limited to £30 consecutive days 2. Maximal dose (prednisone-equivalent) does not exceed 225 mg (5 mg/day for 30 days) 3. Illness was acute in nature and not expected to recur during the remaining treatment period of the study
* Inhaled corticosteroids. At a dose <1200 mg/day beclomethasone equivalent
* Intra-articular injections. A single intra-articular injection allowed every 6 months if the dose of corticosteroid injected is less than an equivalent dose of prednisone 40 mg suspension
* Phenytoin. No phenytoin exposure allowed within 5 years of Month 0 of TOP. Allowed if last phenytoin exposure was >15 years prior to screening for TOP or was between 5-15 years before screening for TOP and for <2 months duration
* Provera® (medroxyprogesterone). Allowed if used according to the label

Laboratory Values and Physical Examination Findings - For excluded laboratory values, the levels shown in the following table are the upper limits for exclusions based on specific test results, with the exception of calculated creatinine clearance and serum 25(OH) vitamin D, for which the limits are lower. All exclusionary laboratory results should be confirmed by a repeat test. Subjects may be excluded for any other clinically abnormal value, as determined by the investigator.

* Fasting serum total calcium (Ca). Subject excluded if value* >10.2 mg/dL**,***
* 24-hour urinary Ca. Subject excluded if value* >360 mg/day**
* Serum total alkaline phosphatase. Subject excluded if value* 3X upper limit of normal for laboratory
* Serum PTH***. Subject excluded if value* >50 pg/mL
* Calculated creatinine clearance*** Subject excluded if value* <50 mL/minute
* Serum 25(OH) vitamin D***. Subject excluded if value* <20 ng/mL

(*)Exclude subject only if repeat assessment confirms the result.

(**)Not to be used as a reason for premature discontinuation during the study. Subjects with elevated values after enrollment are to be managed by the appropriate algorithm (Appendices 2 and 3).

(***)Not an exclusion criterion in OLES

Substance Abuse-Subjects are excluded for a history of alcohol and/or drug abuse as determined by the investigator.

Compliance-Subjects may be excluded for suspected or confirmed poor compliance in completing clinical trial evaluations and/or questionnaires.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2006-10-27 (Actual); Study Completion 2006-10-27 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety of continued once-daily dosing with 100 mg ALX1-11 in postmenopausal osteoporotic women who participated in TOP and OLES clinical trials. | Throughout the study period of approximately 18 months.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the continued efficacy of once-daily treatment with ALX1-11 for maintaining increases in bone mineral density (BMD). | Throughout the study period of approximately 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (9):
  - 'Osteoporosis Medical Center, Beverly Hills, California
  - 'The University of Chicago, Chicago, Illinois
  - 'Michigan Bone & Mineral Clinic, Detroit, Michigan
  - 'Odyssey Research Services, Bismarck, North Dakota
  - Michael J. Lillestol, Fargo, North Dakota
  - 'Odyssey Research Services, Minot, North Dakota
  - 'Rapid City Medical Center, Rapid City, South Dakota
  - 'Brown Clinic, Watertown, South Dakota
  - 'Fletcher Allan Health Center, UHC Campus 1, Burlington, Vermont
- Argentina (3):
  - 'IDIM, Buenos Aires, BUE
  - 'Centro Médico T.I.E.M.P.O, Buenos Aires, BUE
  - 'Centro de Osteopatias Medicas, Capital Federal, CBA

REFERENCES:
- [Derived] Zanchetta JR, Bogado CE, Cisari C, Aslanidis S, Greisen H, Fox J, Lems W. Treatment of postmenopausal women with osteoporosis with PTH(1-84) for 36 months: treatment extension study. Curr Med Res Opin. 2010 Nov;26(11):2627-33. doi: 10.1185/03007995.2010.524121. Epub 2010 Oct 5. PMID 20923256